CLINICAL TRIAL: NCT06550050
Title: Clinical and Molecular Features of Oral Premalignancy and Oral Cancer Associated With Tumor Initiation, Aggressive Behavior, Treatment Response, and Survival Outcomes
Brief Title: Clinical and Molecular Features of Oral Premalignancy and Oral Cancer
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0307; NCI-2024-06602 (Other: NIH-NCI)
Record Dates: First submitted 2024-08-01; First posted 2024-08-12 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms | interventions — Radiation; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinical and molecular features of oral premalignancy and oral cancer
  Interventions: Behavioral: Radiation

INTERVENTIONS:
Behavioral: Radiation — Standard of care
  Other Names: Chemotherapy

SUMMARY:
Investigators will employ serial assessments of tissue biopsy and additional biomarkers that reflect burden of disease and predict treatment response. Patients enrolled on this study will be given the option to provide biological samples before, during, and after treatment, as well as functional outcomes of treatment response. These samples will be utilized to develop and validate prognostic and predictive biomarkers for patients undergoing targeted therapy, immunotherapy, surgery, chemotherapy, and/or radiotherapy.

DETAILED DESCRIPTION:
Primary objectives: Current primary objectives need revision as they focus on diabetes which is not the focus of this study.

* Investigators will examine the role of clinical, environmental, and genetic factors in increasing the risk of developing oral cancers and aggressive oral cancers.
* To identify important environmental and clinical factors contributing to the risk of developing oral cancer or cancer progression
* To identify genetic and molecular factors which contribute to increased risk of developing oral cancers through analysis of germline and somatic genetic alterations
* Investigators will identify clinical and molecular predictors of diagnosis, treatment response, toxicity, and outcomes in patients with oral tumors.
* To identify and validate clinical and molecular prognostic markers that may predict a patient's response to treatment
* To identify and validate clinical and molecular prognostic markers that may predict a patient's risk of developing toxicity related to various modalities of treatment including but not limited to: targeted therapy, chemotherapy, radiation, surgery, and immunotherapy
* To identify and validate clinical and molecular prognostic markers that may predict a patient's prognosis
* To determine whether clinical and treatment factors influence patients' quality of life as assessed by validated self-report instruments routinely incorporated into clinical care pathways
* To identify and validate molecular markers that may improve the diagnosis of oral premalignant or malignant tumors
* To characterize acute and long-term function and quality of life after curative treatment(s)

ELIGIBILITY:
* Aged 18 or older, with a diagnosis of oral premalignant or malignant tumors (eligible diagnoses listed below) or presenting with suspected premalignant or malignant tumors for definitive diagnosis
* Must be able to provide informed consent
* Oral premalignant or malignant tumors presenting for evaluation for the first time at UT MD Anderson Cancer Center
* Oral premalignant or malignant tumors who were previously treated or evaluated at UT MD Anderson Cancer Center who presents for evaluation of progressive or recurrent disease. Newly collected biospecimens and tissue samples will be linked to applicable samples previously collected and banked/stored under PA17-0050, LAB02-427, Lab02-039 and Lab08-0848.

Eligible diagnoses include:

* Leukoplakia
* Erythroplakia
* Mild dysplasia
* Moderate dysplasia
* Severe dysplasia
* Carcinoma in situ
* Squamous cell carcinoma

Exclusion:

- Pregnant women and/or cognitively-impaired adults are excluded from this study.

Exclusion Criteria:

- Prior oral squamous cell carcinoma (OSCC) surgery or OSCC radiation treatment at a non-MDA institution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2064-12-31 (Estimated); Study Completion 2066-12-31 (Estimated)

PRIMARY OUTCOMES:
MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN) | up to 5 years
  The MDASI-HN is a patient-reported outcome questionnaire designed to measure the severity or burden of systemic and head- and neck-specific symptoms and their interference with or effect on patients' daily functioning (Rosenthal, Mendoza et al. 2007, Cleeland 2016). This 28-item multi-symptom inventory is rated according to the last 24 hours at their worst, with 0 being symptoms not present and 10 being as bad as the patient can imagine. Cronbach alpha reliability ranges from 0.72 to 0.92.

SECONDARY OUTCOMES:
M.D. Anderson Dysphagia Inventory (MDADI) | up to 5 years
  The M.D. Anderson Dysphagia Inventory (MDADI) is a written questionnaire to evaluate dysphagia-specific QOL in head and neck cancer patients (Chen, Frankowski et al. 2001). Dysphagia (swallowing difficulty) is a top priority of HNC survivors and a driver of QOL after treatment. The 20-item MDADI questionnaire quantifies an individual's global, physical, emotional, and functional perceptions of his or her swallowing ability. In an internal validation in 100 patients with HNC, concurrent validity was found to be moderate by comparison with the Performance Status Scale (Spearman correlation, 0.47-0.61). Correlation with the physical functional subscale (Spearman correlation, 0.40) and emotional subscale of SF-36 (Spearman correlation, 0.36) demonstrated convergent and divergent validity, respectively, of the MDADI. Test-retest reliability (physical, 0.86; emotional, 0.88; functional, 0.88) and international consistency reliability (overall Cronbach's alpha, 0.96) were sound.

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org